CLINICAL TRIAL: NCT00289458
Title: The Effect of Aquatic Exercise and Aquatic Exercise Combined With Education and Efficacy Enhancement on Improving Indices of Fall Risk in Older Adults With Hip Osteoarthritis: a Randomized Controlled Clinical Trial
Brief Title: Aquatic Exercise and Efficacy Enhancement to Decrease Fall Risk in Older Adults With Hip Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Robert Faulkner Professor, Kinesiology and Cathy Arnold (PhD candidate, Kinesiology) and Associate Professor, School of Physical Therapy, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-REB 05-158
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-07

CONDITIONS: Arthritis
Keywords: older adults, falls, arthritis, aquatic, exercise
MeSH Terms: conditions — Arthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Aquatic Education (Experimental): Exercise combined with education
  Interventions: Behavioral: 2
- Aquatic (Experimental)
  Interventions: Behavioral: exercise
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: exercise — A community aquatic exercise program designed for older adults to improve balance, strength and mobility to decrease the risk of falls.
  Arms: Aquatic
Behavioral: 2 — Same as 1 with the addition of a 1/week educational group program to improve confidence in movement, learn about fall risk and fall prevention and the rationale for the exercises to decrease fall risk.
  Arms: Aquatic Education
Behavioral: Control — no exercise
  Arms: Control

SUMMARY:
The objective of this project is to determine the effect of aquatic exercise and aquatic exercise combined with an education program on decreasing fall risk in older adults with hip osteoarthritis. The hypothesis is that aquatic exercise will improve function, strength and balance and the addition of the education session will enhance confidence in movement.

DETAILED DESCRIPTION:
Older adults with hip osteoarthritis (OA) often experience pain and loss of mobility that significantly impairs their ability to walk, climb stairs, shop or participate in exercise programs. This can result in social isolation, depression and loss of confidence in their ability to manage independently in the community. A decline in physical and psycho-social function leads to increased risk of falling. It is crucial to identify high-risk fallers as well as the best interventions to decrease that risk; hip fractures from falls are devastating, resulting in death or admission to long-term care for the majority who sustain them.

Exercise programs designed to improve balance, strength and mobility can help to improve function and decrease risk of falling. However, individuals with hip OA may have difficulty participating in these programs due to pain. Aquatic exercise offers an activity alternative to improve mobility, strength and decrease fall risk. As well, the addition of a group program designed to enhance confidence in movement may further reduce the risk of falls by improving independence to be more active at home and in the community.

This project will evaluate the effect of aquatic exercise and aquatic exercise combined with a group educational program on decreasing fall risk in older adults with hip OA. Determining optimal fall prevention programs may avert death and loss of quality of life for older adults, clearly an important contribution to preventative health care.

ELIGIBILITY:
Inclusion Criteria:

* over age 65
* clinical diagnosis of hip osteoarthritis

Exclusion Criteria:

* medical condition tha significantly decreases functional ability such that not safe to exercise in a community program
* already exercising in a moderate exercise program 2/week or more

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy M Arnold, MSc, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, Saskatoon, Saskatchewan, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Sept 2005 to 2006, posters in physician offices, senior housing, recreational facilities and advertisements in local newspaper
Groups:
- Control Group: Continued with usual activity and care, no intervention
- Aquatic Exercise: Attended twice per week community aquatic exercise class focussed on improving strength, balance and mobility
- Aquatic Exercise Plus Education: Attended twice per week community aquatic exercise class designed to improve strength, balance, and mobility plus an additional educational class once per week to learn about fall risk, and improve confidence in ability to prevent falls.
Period: Overall Study
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Started | 25 | 26 | 28
Completed | 19 | 20 | 22
Not Completed | 6 | 6 | 6
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 3 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education | Total
Number analyzed (Participants) | 25 | 26 | 28 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 25 | 26 | 28 | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 75.8 (6.2) | 74.4 (7.5) | 73.2 (4.8) | 74.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 20 | 56
  Male | 9 | 6 | 8 | 23
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 26 | 28 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change in Balance
Description: Berg Balance Scale range 0 - 36 (36 is excellent balance, 0 is poor or no ability for standing balance)
Time Frame: baseline and 11 weeks
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
units on a scale | 0.2 (2.3) | 1.2 (2.3) | 1.0 (3.5)

2. Primary Outcome: Change in Chair Stands
Description: change in number of repetitions (the number of times moving from full sitting to full standing in 30 seconds)
Time Frame: baseline and 11 weeks
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: number of stands per 30 seconds
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
number of stands per 30 seconds | 0.6 (1.7) | 0.6 (1.7) | 1.5 (2.0)

3. Primary Outcome: Change in Walking
Description: change in 6 minute walk (distance in meters covered in 6 minutes)over 11 weeks
Time Frame: baseline and 11 weeks
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: unit of scale (meters per 6 minutes)
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
unit of scale (meters per 6 minutes) | 0.3 (70.7) | 14.5 (70.3) | 43.3 (63.8)

4. Primary Outcome: Change in Falls-Efficacy
Description: change in Activities Balance Confidence Scale (0 - 100, 100 represents high confidence, 0 represents low confidence)
Time Frame: baseline and 11 weeks
Population: ITT and LOCF
Measure: Mean (Standard Deviation); unit: unit of scale
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
unit of scale | 2.4 (10.7) | 0.8 (21.1) | 5.8 (12.4)

5. Secondary Outcome: Change in Physical Activity
Description: change in Physical Activity Scale for the Elderly (0 - up to 300, higher score more active)
Time Frame: baseline and 11 weeks
Measure: Mean (Standard Deviation); unit: unit of scale
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
unit of scale | 101.4 (47.3) | 106.9 (50.4) | 96.6 (32.7)

6. Primary Outcome: Change in Dual Task Function
Description: change in Timed Up and Go Cognitive Test (time in sec., lower number means better performance)
Time Frame: baseline and 11 weeks
Measure: Mean (Standard Deviation); unit: unit of scale (seconds)
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Number analyzed (Participants) | 25 | 26 | 28
unit of scale (seconds) | 0.2 (4.3) | 0.7 (3.1) | 2.5 (5.1)

ADVERSE EVENTS:
Arm/Group | Control Group | Aquatic Exercise | Aquatic Exercise Plus Education
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes